CLINICAL TRIAL: NCT01279863
Title: Vibration Response Imaging (VRI) in Children With Acute Respiratory Symptoms.
Brief Title: VRI in Children With Acute Respiratory Symptoms.
Acronym: VRI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Liora Kornreich, MD, Schneider children's Medical center of Israel
Other Study IDs: 5500-DB048
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2010-05

CONDITIONS: Pneumonia; Fever
Keywords: Pneumonia; Cough; Shortness of breath; VRI
MeSH Terms: conditions — Pneumonia; Fever; Cough; Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The VRI technology provides a radiation free dynamic image of the lung, by using a combination of well-known technologies, i.e. acoustic sensors, and a proprietary algorithm. The aim of the study is to determine if the VRI examination may contribute to the diagnosis and follow up of pneumonia in children, and therefore reduce the number of chest radiographs and the exposure to ionizing radiation. Children referred by ED for chest x-ray,for the evaluation of pneumonia, will undergo VRI as well. The two modalities will be read independently and then the findings will be compared, in order to asses the potential role of the VRI to the management of pneumonia in children.

DETAILED DESCRIPTION:
Background Several widely used imaging modalities are available today for the human lung. Conventional radiology, CT, and to a lesser extent MRI, as well as nuclear medicine in some indications are well established and most commonly used. Methods using acoustic signals, most notably ultrasound, have not been successfully developed. This is primarily due to the fact that the acoustic damping of the lung parenchyma is prohibitively high at high frequencies .

Assessment of alterations in the structure and function of thoracic organs that occur in disease often gives rise to measurable changes in lung sound production and transmission. Acoustic assessment with a stethoscope is a commonly used method to assess these structural and functional changes. However, auscultation with a stethoscope has many limitations. It is a subjective process that depends on the individual's own hearing, experience and ability to differentiate between different sound patterns. In addition, quantitative measurements and documentation are not easy to be produced. Moreover, the stethoscope has a frequency response that attenuates frequency components of the lung sound signal above 120Hz, and the human ear is not very sensitive to the lower frequency band.

Analysis of acoustic sounds by computer is more likely to be successful in clinical applications when it is based on mathematical models of the underlying physical mechanisms of respiratory sound production. Such models allow for the interaction of mechanical forces, airflow and sound transmission within the respiratory tract to be understood and related to the different disease processes.

The VRI technology, to the best of our knowledge, is the first of its kind to provide a radiation free dynamic image of the lung, by using a combination of well-known technologies, i.e. acoustic sensors, and a proprietary algorithm.

Since the acoustic response of a body depends on its structural properties, complex structures can exhibit acoustic responses, which may vary in space, time and frequency. Moreover, any structural alteration, such as a bronchial obstruction or space occupying infiltration, is reflected by a corresponding modification of the acoustic response.

The VRI takes advantage of this physical principle, by means of an imaging system. By attaching a two dimensional matrix of acoustic transducers to the back of the patient, a dynamic image that integrates the acoustic characteristics of the underlying structure is generated.

The VRI device may provide a complementary diagnostic tool for lung examination and aid the physician in determining whether a chest x-ray should be performed.

Study Device The VRI system is a computerized-based, radiation free device intended for non-invasive recording, audio reproduction, and dynamic image display of vibration response to the airflow during respiration. (The VRI system incorporates a flow volume sensor in which the patient may/may not breathe through it). The VRI system incorporates pressure sensors (electronic stethoscopes) that have been specially adapted to capture and record the energy created by the airflow in the lungs during the respiration process. Sensors are mounted in two sensor matrices, which are attached to the patient's back by a low vacuum and/or biocompatible medical stickers method. The signals are transmitted through wires from the sensor matrix to the hardware board. The analog signals are then processed online on a multi-channels hardware board by amplifying, sampling and A/D conversion. The digital data is transmitted to the PC platform. Once on the PC platform, Deep Breeze proprietary algorithms generate the dynamic lung image.

Risk Analysis Unlike X-Ray based methodologies, which expose the subject to ionization radiation, the VRI is radiation free.

The VRI elements that come into contact with the subject's skin are biocompatible.

The VRI has been approved by an independent authorized laboratory to be electrically safe.

In addition, so far, no adverse events, risks of illness, injuries, or discomforts have been associated with the use of the VRI in previous studies. Therefore, it is reasonable to conclude that the VRI does not pose any risk to the subjects and/or operators.

Study Rationale Various reports and studies have suggested that a reduction of up to 50% of X rays could be achieved without detriment to the care and treatment of patients. A considerable number of the X-ray procedures carried out today produce no meaningful or useful diagnostic information and it is the elimination of these examinations that would bring about this reduction, as stated by the Irish Institute of Radiography.

One study investigated the use of the chest X-ray (CXR) in a typical urban practice with reference to the Royal College of Radiology (RCR) guidelines. A total of 569 CXRs were performed in 482 patients. Thirty per cent of the CXRs were assessed as being "not indicated" and a significant percentage of requests did not come within the RCR guidelines.

According to the Royal College of Radiologists (RCR) Working Party at least 20% of the radiological examinations carried out in NHS hospitals are clinically unhelpful. This translates over the whole country to an annual total of 7 million unnecessary X-ray examinations costing about £60 million, with the highest numbers of unnecessary X-ray examinations being those of chest and the greatest financial costs arising from examinations of the chest and from barium investigations. , , Unnecessary radiation exposure during medical procedures should be avoided. This is particularly important when the patient is a child, since children exposed to radiation are at a relatively greater risk than adults. The American College of Radiology has noted, "Because they have more rapidly dividing cells than adults and have longer life expectancy, the odds that children will develop cancers from x-ray radiation may be significantly higher than adults." It has been estimated by the National Research Council's Committee on the Biological Effects of Ionizing Radiation that children less than 10 years of age are several times more sensitive to radiation than middle-aged adults .

The VRI device may provide a complementary diagnostic tool for lung examination and aid the physician in determining whether a chest x-ray (CXR) is necessary and thereby reduce the number of negative CXR.

Summary of Clinical Experience The device has already been used for investigational purposes in a number of medical centers (Israel, USA, Europe and Japan). All clinical studies were performed in accordance with the ICH-GCP guidelines as well as the local laws and regulations relevant to the use of new diagnostic devices.

Recorded data was collected and analyzed for more than 3000 adult subjects during a period of more than three years. No related adverse events were reported during the studies.

Study Objective

* The principal objective of the pilot study is to acquire database of pneumonia cases in children.
* The secondary objective is to correlate the clinical and CXR data with the VRI results.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be entered into the study:

1. Subject's parent or legal guardian, is able and willing to read the Informed Consent, understands the Informed Consent, and provides written Informed Consent for the subject; if the minor child is in fact able to give consent, the minor's consent must be obtained in addition to the consent of the minor's legal guardian.
2. Boy or girl in the age range of 3-18 years.
3. Patient presented with acute respiratory complaints, acute cough, onset of shortness of breath, or fever.
4. Patient referred by ED physician and presented for CXR.

Exclusion Criteria:

Any of the following will exclude the patient from study:

1. Body habitus or skin condition that might prevent the placement of the sound sensors on the back (e.g. severe scoliosis, kyphosis, chest wall deformation, skin lesion on the back or compression fracture);
2. Potentially contagious skin lesion on the back;

4. Subject has had lung surgery; 5. Subject was prescribed the CXR for monitoring or follow up of a lung condition that pre-existed the current, acute symptoms.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, 3-18 years old
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-08 (Estimated); Study Completion 2012-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Liora Kornreich, MD, Principal Investigator — Schneider Children's Medical Center, Israel; Gadi Horev, MD, Study Chair — Schneider Children's Medical Center, Israel; Michael Schwarz, MD, Study Chair — Schneider Children's Medical Center, Israel; Osnat Konen, MD, Study Chair — Schneider Children's Medical Center, Israel; Nadine Berkowitz, MD, Study Chair — Schneider Children's Medical Center, Israel; Yehezkel Waisman, MD, Study Chair — Schneider Children's Medical Center, Israel
Locations (1):
- Schneider medical center of Israel, Imaging Department, Petah Tikva, Israel